CLINICAL TRIAL: NCT00423826
Title: A Pilot Study of Double Cord Blood Stem Cell Transplantation in Patients With Hematologic Malignancies
Brief Title: Umbilical Cord Blood Stem Cell Transplant in Treating Patients With Hematologic Cancer or Other Disease
Status: No longer available | Type: Expanded Access
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Voravit Ratanatharathorn, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Other Study IDs: CDR0000518230; P30CA022453 (NIH); WSU-2006-059 (Other: Barbara Ann Karmanos Cancer Institute); WSU-112506MP2F (Other: Wayne State University Institutional Review Board)
Record Dates: First submitted 2007-01-16; First posted 2007-01-18 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-02

CONDITIONS: Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Precancerous Condition; Secondary Myelofibrosis
Keywords: accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; childhood chronic myelogenous leukemia; relapsing chronic myelogenous leukemia; adult acute lymphoblastic leukemia in remission; recurrent adult acute lymphoblastic leukemia; childhood acute lymphoblastic leukemia in remission; recurrent childhood acute lymphoblastic leukemia; adult acute myeloid leukemia in remission; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); recurrent adult acute myeloid leukemia; adult acute minimally differentiated myeloid leukemia (M0); adult acute myeloblastic leukemia without maturation (M1); adult acute myeloblastic leukemia with maturation (M2); adult acute promyelocytic leukemia (M3); adult acute myelomonocytic leukemia (M4); adult acute monoblastic leukemia (M5a); adult acute monocytic leukemia (M5b); adult erythroleukemia (M6a); adult pure erythroid leukemia (M6b); adult acute megakaryoblastic leukemia (M7); childhood acute myeloblastic leukemia without maturation (M1); childhood acute myeloblastic leukemia with maturation (M2); childhood acute promyelocytic leukemia (M3); childhood acute myelomonocytic leukemia (M4); childhood acute monoblastic leukemia (M5a); childhood acute monocytic leukemia (M5b); childhood acute erythroleukemia (M6); childhood acute megakaryocytic leukemia (M7); childhood acute myeloid leukemia in remission; secondary myelodysplastic syndromes; recurrent childhood acute myeloid leukemia; refractory chronic lymphocytic leukemia; recurrent adult Hodgkin lymphoma; recurrent/refractory childhood Hodgkin lymphoma; adult grade III lymphomatoid granulomatosis; adult nasal type extranodal NK/T-cell lymphoma; Waldenstrom macroglobulinemia; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; recurrent marginal zone lymphoma; secondary acute myeloid leukemia; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; extramedullary plasmacytoma; isolated plasmacytoma of bone; monoclonal gammopathy of undetermined significance; primary systemic amyloidosis; refractory multiple myeloma; de novo myelodysplastic syndromes; childhood acute minimally differentiated myeloid leukemia (M0); childhood grade III lymphomatoid granulomatosis; childhood nasal type extranodal NK/T-cell lymphoma; recurrent adult grade III lymphomatoid granulomatosis; recurrent childhood large cell lymphoma; recurrent childhood lymphoblastic lymphoma; childhood diffuse large cell lymphoma; childhood immunoblastic large cell lymphoma; Burkitt lymphoma; recurrent childhood small noncleaved cell lymphoma; previously treated myelodysplastic syndromes; splenic marginal zone lymphoma; recurrent childhood grade III lymphomatoid granulomatosis; recurrent adult lymphoblastic lymphoma; recurrent small lymphocytic lymphoma; secondary myelofibrosis
MeSH Terms: conditions — Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Precancerous Conditions; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Congenital Abnormalities; Leukemia, Myeloid, Acute; Leukemia, Promyelocytic, Acute; Leukemia, Myelomonocytic, Acute; Leukemia, Monocytic, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Lymphocytic, Chronic, B-Cell; Hodgkin Disease; Recurrence; Lymphoma, Extranodal NK-T-Cell; Waldenstrom Macroglobulinemia; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Monoclonal Gammopathy of Undetermined Significance; Immunoglobulin Light-chain Amyloidosis; Dendritic Cell Sarcoma, Interdigitating | interventions — Busulfan; Cytarabine; fludarabine phosphate; Mycophenolic Acid; Tacrolimus; Cord Blood Stem Cell Transplantation; Whole-Body Irradiation

INTERVENTIONS:
Drug: Busulfan — 3 mg/kg intravenously over 3 hours
  Other Names: Busulfex®; Myleran®
Drug: Cytarabine — Patients with previous history of CNS involvement will receive pre-transplant intrathecal Cytarabine (Ara-C) (30 mg/M2) therapy.
  Other Names: DepoCyt(TM); Liposomal Ara-C
Drug: Fludarabine phosphate — 25 mg/M2/day IV
  Other Names: Fludara
Drug: mycophenolate mofetil — Orally at the dose of 1 gm every 8 hours.
  Other Names: Cellcept
Drug: tacrolimus — 0.015 mg/kg IV every 12 hours by continuous infusion.
  Other Names: Advagraf; Prograf; Protopic
Procedure: allogeneic hematopoietic stem cell transplantation — 10 days post drug intervention
Procedure: umbilical cord blood transplantation — 10 days post drug intervention
Radiation: total-body irradiation — 10 days post drug intervention

SUMMARY:
RATIONALE: Giving low doses of chemotherapy and total-body irradiation before a donor umbilical cord blood stem cell transplant helps stop the growth of cancer or abnormal cells. It also stops the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune cells and help destroy any remaining cancer or abnormal cells (graft-versus-tumor effect). Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving tacrolimus and mycophenolate mofetil before the transplant may stop this from happening.

PURPOSE: This clinical trial is studying how well umbilical cord blood stem cell transplant works in treating patients with hematologic cancer or other disease.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy of double umbilical cord blood stem cell transplantation using a conditioning regimen comprising lower doses of busulfan and fludarabine phosphate and low-dose total body irradiation, in terms of stem cell engraftment at 60 days post transplantation, in patients with hematologic cancer or other diseases.
* Determine the merits of conducting a larger, comparative study of this regimen.

Secondary

* Determine mortality within 100 days of transplantation in these patients.

OUTLINE: This is a pilot study.

* Reduced-intensity conditioning regimen: Patients receive busulfan IV over 3 hours on days -9 to -8 and fludarabine phosphate IV on days -7 to -3. Patients then undergo low-dose total body irradiation on day 0.
* Graft-versus-host disease prophylaxis: Patients receive tacrolimus IV twice daily and mycophenolate orally or IV three times daily beginning on day -3.
* CNS prophylaxis and/or treatment: Patients with a history of CNS involvement receive prophylactic cytarabine (Ara-C) intrathecally (IT) prior to transplant. Patients also undergo lumbar puncture (LP) to test for active CNS disease. Patients with cerebrospinal fluid positive for leukemia receive Ara-C IT every 2-3 days until a repeat LP shows no remaining leukemic cells. Three days after the last LP and after one final dose of Ara-C, patients begin the conditioning regimen.
* Double umbilical cord blood (UCB) donor stem cell transplantation (SCT): Patients undergo double UCB donor SCT on day 0.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diagnosis of 1 of the following:

  * Acute myeloid leukemia meeting the following criteria:

    * M0-M7 histologic subtypes by French-American-British classification
    * Previously treated disease
    * Meets 1 of the following criteria:

      * Persistent disease as evidenced by 5-30% persistent blasts in bone marrow after induction or salvage therapy
      * In second or subsequent complete remission (CR)
      * In first CR with 1 of the following high-risk features:

        * Philadelphia chromosome present
        * Noncore-binding factor type of chromosomal abnormalities
  * Myelodysplastic syndromes with 1 of the following International Prognostic Scoring System (IPSS) scores:

    * Intermediate-1
    * Intermediate-2
    * High-risk score with transfusion dependence
  * Chronic myelogenous leukemia meeting 1 of the following criteria:

    * In accelerated or blastic phase
    * Failed prior imatinib mesylate therapy
  * Acute lymphoblastic leukemia meeting 1 of the following criteria:

    * In first CR with any of the following high-risk features:

      * Philadelphia chromosome present
      * Translocation t(4;11) present
      * WBC > 30,000/mm³ (adult patients)
      * More than 4 weeks from initiation of treatment was required to achieve CR (adult patients)
      * DNA index of near haploid (N=23 chromosomes) (pediatric patients)
    * In second or subsequent CR
    * Persistent disease as evidenced by 5-20% persistent blasts in bone marrow after induction or salvage therapy
  * Hodgkin's or non-Hodgkin's lymphoma meeting the following criteria:

    * Recurrent or refractory disease
    * Tumor ≤ 5 cm in diameter
  * Myeloma or plasma cell neoplasm meeting 1 of the following staging criteria:

    * Stage III at presentation
    * Stage I-II at presentation

      * Not responding OR progressed after first-line therapy
  * Chronic lymphocytic leukemia or Waldenstrom's macroglobulinemia with refractory or progressive disease after first-line therapy
* No 5-6/6 HLA-matched related or 7-8/8 HLA-matched unrelated marrow or peripheral blood stem cell donor available
* No single 4-6/6 HLA-A, -B, or -DRB1-matched umbilical cord blood unit ≥ 3.5 x 10^7 nucleated cells/kg available

PATIENT CHARACTERISTICS:

* ECOG performance status (PS) 0-2 OR Karnofsky or Lansky PS 70-100%
* Not pregnant
* Fertile patients must use effective contraception prior to and during study participation
* HIV negative
* Bilirubin < 3.0 mg/dL
* AST and ALT ≤ 3 times upper limit of normal
* Creatinine < 2.0 mg/dL OR creatinine clearance > 50 mL/min
* Cardiac ejection fraction > 50% by echocardiogram OR shortening fraction > 27%
* No uncontrolled symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* FEV_1 > 50% of normal
* Forced vital capacity > 50% of normal
* DLCO normal
* Oxygen saturation > 92% on room air (for patients < 5 years of age)
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to busulfan and fludarabine phosphate
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance
* No other uncontrolled illness

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 4 weeks since prior and no concurrent surgery
* At least 4 weeks since prior and no other concurrent investigational or commercial agents or therapies for the malignancy, including chemotherapy, biologic therapy, or radiotherapy

Max Age: 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2007-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Voravit Ratanatharathorn, MD, Study Chair — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States